CLINICAL TRIAL: NCT06100081
Title: Real-time Targeted Fluorescence Endoscopy for Detection of the Primary Cancer Lesion in Patients With a Metastasis of Unknown Primary Tumor in the Head and Neck
Acronym: REFLECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10949
Record Dates: First submitted 2023-04-17; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Unknown Primary Tumors; Oropharynx Cancer
MeSH Terms: conditions — Neoplasms, Unknown Primary; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Patients with cancer of unknown primary most probable originating from the head and neck area
  Interventions: Diagnostic Test: Detection of lesions using fluorescence molecular imaging

INTERVENTIONS:
Diagnostic Test: Detection of lesions using fluorescence molecular imaging — Using a fluorescence camera, lesions will be detected and biopsies will be taken to try and find cancer of unknown primary

SUMMARY:
In current diagnostic work-up of patients with a cancer of unknown primary (CUP), approximately 50% of the primary tumor lesions remains undetected. Identification of the primary tumor site results in minimizing the potential morbidity from treatment by reducing morbidity by omitting the need for a mucosectomy of the bilateral base of tongue and tonsils, reducing the radiation field and better oncologic outcome than those with unidentified primary tumor. Clearly, new endoscopic 'real-time' imaging techniques are needed to visualize mucosal changes associated with head and neck squamous cell carcinoma and increase detection rate of the primary tumor. Targeted fluorescence endoscopy enables the visualization of targeted tumor-specific biomarkers by using fluorescence, thereby enhancing the contrast between normal mucosa and tumor tissue. This could improve the detection of the primary tumor in cases where the primary tumor is not detected with white light endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Cytology and/or histology-confirmed diagnosis of squamous cell carcinoma most likely originating from the head & neck area and scheduled to undergo endoscopy of the upper aerodigestive tract as decided by the multidisciplinary head and neck tumor board of the UMCG;
* The primary tumor was not identified during standard diagnostic work-up in the outpatient clinic including physical head and neck examination, fiberoptic laryngoscopy, chest X-ray, CT and PET/CT;
* Age ≥ 18 years;
* Written informed consent;

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent;
* Concurrent uncontrolled medical conditions;
* Received an investigational drug within 30 days prior to the dose of cetuximab-800CW;
* History of myocardial infarction, cerebrovascular accident, uncontrolled cardiac heart failure, significant liver disease (ALT >3X upper limits of normal or increased total bilirubin) or unstable angina within 6 months prior to enrollment;
* Inadequately controlled hypertension with or without current antihypertensive medications;
* History of allergy or infusion reactions cetuximab or other monoclonal antibody therapies;
* Pregnant or lactating women. Documentation of a negative pregnancy test must be available for women of childbearing potential. Moreover, the need to be willing to ensure that she or her partner uses effective contraception during the trial and for 6 months thereafter. Woman of childbearing potential are premenopausal women with intact reproductive organs and women less than two years after menopause;
* Evidence of QT prolongation on pretreatment ECG (greater than 440 ms in males or greater than 450 ms in females)
* Patients receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
* Life expectancy < 12 weeks;
* Karnofsky performance status < 70%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy in detecting primary tumours compared to white light endoscopy. | During surgery
  To determine the feasibility of targeted fluorescence endoscopy compared to white light endoscopy and a mucosectomy using cetuximab-800CW for the detection of the primary tumor in patients with CUP

SECONDARY OUTCOMES:
Safety aspects of cetuximab-800CW | through study completion
  To obtain information on safety aspects of cetuximab-800CW administration by registration of side effects, adverse events (AE), serious adverse events (SAE) and suspected unexpected serious adverse reactions (SUSAR);
Accuracy in detecting primary tumours with flexible fluorescence laryngoscopy at the outpatient clinic for primary tumor detection rates | Flexible endoscopy will be performed 1-0 days before surgery.
  Accuracy in detecting primary tumours with flexible fluorescence laryngoscopy at the outpatient clinic for primary tumor detection rates
To quantify intrinsic fluorescence signals of cetuximab-800CW; | During the procedure
  To quantify intrinsic fluorescence signals of cetuximab-800CW;
To determine if ex vivo fluorescence imaging using cetuximab-800CW can be used for assessment of the surgical specimen after mucosectomy; | immediatly after the procedure
  To determine if ex vivo fluorescence imaging using cetuximab-800CW can be used for assessment of the surgical specimen after mucosectomy;
To determine the specificity and positive predictive value of TFE and WLE for the detection of the primary tumor in patients with CUP. | end of study
  To determine the specificity and positive predictive value of TFE and WLE for the detection of the primary tumor in patients with CUP.
To correlate and validate fluorescence signals in vivo and ex vivo with histopathology. | 1-2 weeks after procedure
  To correlate and validate fluorescence signals in vivo and ex vivo with histopathology.
To study health-related quality of life data regarding the standard of care mucosectomy procedures performed with transoral robot surgery using the QLQ-C30, QLQH&N35 en de SWAL-QoL. | up to 6 weeks after surgery
  To study health-related quality of life data regarding the standard of care mucosectomy procedures performed with transoral robot surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided